CLINICAL TRIAL: NCT00229177
Title: Controlled Study of ONO-2506 in Patients With Acute Ischemic Stroke
Brief Title: Study of ONO-2506 in Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-2506-08
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Stroke
Keywords: ONO-2506; stroke; Acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — ONO2506

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- P (Placebo Comparator)
  Interventions: Drug: ONO-2506
- E1 (Experimental)
  Interventions: Drug: ONO-2506
- E2 (Experimental)
  Interventions: Drug: ONO-2506

INTERVENTIONS:
Drug: ONO-2506 — Once daily one-hour intravenous infusion at 12/mg/kg/hr for 7 days
  Arms: E2
Drug: ONO-2506 — Once daily one-hour intravenous infusion at 0 mg/kg/hr for 7 days
  Arms: P
Drug: ONO-2506 — Once daily one-hour intravenous infusion at 8 mg/kg/hr for 7 days
  Arms: E1

SUMMARY:
The purpose of this study is to determine the efficacy and safety of ONO-2506 compared to placebo in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have a clinical diagnosis of acute ischemic stroke
2. Subjects within 72 hours after onset of the stroke
3. Other inclusion criteria may apply.

Exclusion Criteria:

1. Subjects who are scheduled to have surgical operations likely to affect the prognosis (including intravascular surgery and circulatory reconstruction)
2. Subjects who are pregnant or lactating, or who have child-bearing potential, or who wish to become pregnant.
3. Other exclusion criteria may apply.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale at 90 days | 90 days

SECONDARY OUTCOMES:
Modified Rankin Scale at 30 days | 30 days
National Institutes of Health Stroke Scale (NIHSS), Barthel Index (BI), and Glasgow Outcome Scale (GOS) at 90 days | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - Chugoku Region Facility, Chugoku
  - Chubu Region Facility, Chūbu
  - Hokkaido Region Facility, Hokkaido
  - Hokuriku Region Facility, Hokuriku
  - Kanto Region Facility, Kanto
  - Kinki Region Facility, Kinki
  - Kyushu Region Facility, Kyushu
  - Shikoku Region Facility, Shikoku
  - Tohoku Region Facility, Tohuku